CLINICAL TRIAL: NCT03476395
Title: Evaluation of Sport Specific Adaptations and Risk Factors at the Shoulder Joint and Core Stability Among Female Volleyball Players With and Without Overuse Related Shoulder Symptoms
Brief Title: Sport Specific Adaptions in Female Volleyball Players
Status: Completed | Type: Observational
Sponsor: Zurich University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Lydia Bucher, Student, Zurich University of Applied Sciences
Other Study IDs: 2017-00762
Record Dates: First submitted 2017-12-21; First posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Overuse Related Shoulder Problems

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: shoulder range of motion in IR/ER, strength of the IR/ER muscles and Scapular Dyskinesis Test. Core endurance test. — Passive shoulder range of motion using a digital application Clinometer. Isometric strength of the shoulder IR/ER using a HHD measured. Scapular Dyskinesis Test uses a visual scoring system. Core Endurance is teste by measuring the time (s).

SUMMARY:
The shoulder joint is the second most affected body part of all overuse injuries in overhead athletes. Due to the repetitive throwing motion overhead athletes show the following characteristic adaptations of their dominant shoulder: Loss of internal rotation (IR) and gain of external rotation (ER), reduced muscle strength of the shoulder external rotators and scapular dyskinesis. On the one hand these adaptations are normal and necessary for a powerful throwing performance. On the other hand the amount of adaptation seems to play a crucial role in developing overuse symptoms and therefore becoming a risk factor. Most previous studies investigating throwing specific adaptations and risk factors focused on overhead sports like baseball, handball or tennis, whereas similar research in volleyball is still insufficient. Therefore the aim of this study is to evaluate if sport specific adaptations are present in female volleyball players and if yes, if there is a difference of the extent of these adaptations in volleyball players with overuse symptoms and players without.

DETAILED DESCRIPTION:
Background The shoulder joint is the second most affected body part of all overuse injuries in overhead athletes.Prevalence of a history of shoulder problems related to overuse in volleyball players was reported to be approximately 60%. Typical overuse symptoms like pain seriously limit progress in performance and the individual career options of volleyball players.

Due to the repetitive throwing motion overhead athletes show the following characteristic adaptations of their dominant (Ds), compared to the non-dominant (NDs) shoulder: 1) Loss of internal rotation (IR) and gain of external rotation (ER), by preserving the total rotational motion (TROM). 2) Reduced muscle strength of the shoulder external rotators (ER). 3) Scapular dyskinesis. On the one hand these adaptations are normal and necessary for a powerful throwing performance. On the other hand the amount of adaptation seems to play a crucial role in developing overuse symptoms and therefore becoming a risk factor; e.g. loss of IR, also known as glenohumeral internal rotation deficit (GIRD) of more than 20° side difference, and a loss of TROM of the Ds, were defined as risk factors in baseball players. Moreover decreased muscle strength of ER (OR: 0.71 per 10N decrease) in the Ds as well as obvious scapular dyskinesis were associated with increased risk of overuse related shoulder symptoms (ORSS). Nevertheless there are still overhead athletes showing these adaptations or risk factors without being symptomatic.

Recently, several authors underlined the importance of core stability related to the kinetic chain during an overhead throwing task. It is hypothesised that symptomatic athletes may overload the shoulder girdle through altered biomechanics in an effort to compensate for insufficient power generated by the core musculature. The most reliable measurements to asses core stability components are core endurance tests.

Most previous studies investigating throwing specific adaptations and risk factors focused on overhead sports like baseball, handball or tennis, whereas similar research in volleyball is still insufficient. Moreover, no one ever investigated core endurance and its possible association with (ORSS) in volleyball players.

Objective The first aim is, to evaluate if sport specific adaptations such as IR ROM deficit, gain of ER ROM, ER strength deficit, alterations in TROM and scapular dyskinesis are present in female volleyball players and if yes, if there is a difference of the extent of these adaptations in volleyball players with ORSS and players without.

The second aim is, to evaluate if there is a difference in core endurance in volleyball players with ORSS and players without and if there is a correlation of core endurance and shoulder related risk factors such as ER strength deficit and scapular dyskinesis?

ELIGIBILITY:
Inclusion Criteria:

* female
* being member of a Nat. League B/Nat. League A Volleyball Team in season 2017/2018
* minimum age 16 years
* sufficient understanding/speaking of the German language
* signed informed consent

Exclusion Criteria:

* having had any surgery at the shoulder joint of the dominant or non- dominant side within last six month
* having had any self reported trauma at the shoulder joint of the dominant or non-dominant side, which limits training or match participation of more than 50%
* limitation of more than 50% in training or match participation caused by a surgery or trauma at the core or lower extremity

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: female volleyball players from the German part of Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-03-18 (Actual)

PRIMARY OUTCOMES:
isometric strength of shoulder internal and extern rotators | 2017
  Isometric strength is measured in Newton (N) using a digital handheld dynamometer (HHD; Model 01165, Lafayette Instrument Company, USA). The participants are placed in supine with their shoulder in 0° abduction (ABD) a small towel roll is used to maintain the humerus in a neutral position and their elbow flexed to 90°. The forearm is fixed to the core using a fixation band. The HHD is placed on the dorsal or ventral aspect of the forearm for ER and IR, directly proximal to wrist joint line. Players are asked to perform all strength measures twice with a rest of 30 sec. between the two attempts. The mean of the two attempts is recorded.
passive glenohumeral range of motion in internal and external rotation | 2017
  Glenohumeral ROM is measured in degrees (°) on both sides using a digital application Clinometer (Plaincode Software Solutions, Peter Breitling, Stephanskirchen Germany, version 4.5 (1511062) on iOS). Participants are placed supine, the shoulder positioned in 90° of abduction, a small towel roll is used to maintain the position of the humerus in neutral and their elbow is flexed to 90°. A splint is fastened around the forearm, to attach the smartphone. The assessor palpates the coracoid process with the thumb and the spine of the scapula with the fingers to control for scapular movement. The shoulder is passively moved to the end of ROM (EOR) into IR and ER. EOR of IR and ER is defined at the point at which the scapula is moving. The mean of two trials for IR and ER is used for data analysis.
scapular dyskinesis | 2017
  Scapular control is evaluated using the scapular dyskinesis test (SDT). In standing position players held two dumbbells each in one hand. Players are instructed to bilaterally elevate their arms overhead as far as possible to a 3-second count with thumbs positioned upwards and then lower to a 3-second count. Five repetitions are performed while they are visually observed from posterior. The final rating classifies scapula control as normal, subtle abnormal or obvious abnormal.

SECONDARY OUTCOMES:
core stability | 2017
  Core stability is assessed using core endurance tests in seconds (s). Tests are performed in a sit up position in 60° Flexion and in side plank position on both sides. Players are instructed to hold their back and hip to the upright position for as long as possible. The test terminates, when the player is not able to hold the position anymore.

CONTACTS AND LOCATIONS:
Locations (1):
- ZHAW, Winterthur, Switzerland

REFERENCES:
- [Background] Clarsen B, Bahr R, Heymans MW, Engedahl M, Midtsundstad G, Rosenlund L, Thorsen G, Myklebust G. The prevalence and impact of overuse injuries in five Norwegian sports: Application of a new surveillance method. Scand J Med Sci Sports. 2015 Jun;25(3):323-30. doi: 10.1111/sms.12223. Epub 2014 Mar 30. PMID 24684525
- [Background] Ruotolo C, Price E, Panchal A. Loss of total arc of motion in collegiate baseball players. J Shoulder Elbow Surg. 2006 Jan-Feb;15(1):67-71. doi: 10.1016/j.jse.2005.05.006. PMID 16414471
- [Background] Burkhart SS, Morgan CD, Kibler WB. The disabled throwing shoulder: spectrum of pathology Part I: pathoanatomy and biomechanics. Arthroscopy. 2003 Apr;19(4):404-20. doi: 10.1053/jars.2003.50128. PMID 12671624
- [Background] Borsa PA, Laudner KG, Sauers EL. Mobility and stability adaptations in the shoulder of the overhead athlete: a theoretical and evidence-based perspective. Sports Med. 2008;38(1):17-36. doi: 10.2165/00007256-200838010-00003. PMID 18081365
- [Background] Burkhart SS, Morgan CD, Kibler WB. The disabled throwing shoulder: spectrum of pathology Part III: The SICK scapula, scapular dyskinesis, the kinetic chain, and rehabilitation. Arthroscopy. 2003 Jul-Aug;19(6):641-61. doi: 10.1016/s0749-8063(03)00389-x. No abstract available. PMID 12861203
- [Background] Wilk KE, Arrigo CA, Hooks TR, Andrews JR. Rehabilitation of the Overhead Throwing Athlete: There Is More to It Than Just External Rotation/Internal Rotation Strengthening. PM R. 2016 Mar;8(3 Suppl):S78-90. doi: 10.1016/j.pmrj.2015.12.005. PMID 26972270
- [Background] Cools AM, Johansson FR, Borms D, Maenhout A. Prevention of shoulder injuries in overhead athletes: a science-based approach. Braz J Phys Ther. 2015 Sep-Oct;19(5):331-9. doi: 10.1590/bjpt-rbf.2014.0109. Epub 2015 Sep 1. PMID 26537804
- [Background] Kibler WB, Press J, Sciascia A. The role of core stability in athletic function. Sports Med. 2006;36(3):189-98. doi: 10.2165/00007256-200636030-00001. PMID 16526831
- [Background] Reeser JC, Fleisig GS, Bolt B, Ruan M. Upper limb biomechanics during the volleyball serve and spike. Sports Health. 2010 Sep;2(5):368-74. doi: 10.1177/1941738110374624. PMID 23015961
- [Background] Evans K, Refshauge KM, Adams R. Trunk muscle endurance tests: reliability, and gender differences in athletes. J Sci Med Sport. 2007 Dec;10(6):447-55. doi: 10.1016/j.jsams.2006.09.003. Epub 2006 Dec 1. PMID 17141568
- [Background] Myklebust G, Hasslan L, Bahr R, Steffen K. High prevalence of shoulder pain among elite Norwegian female handball players. Scand J Med Sci Sports. 2013 Jun;23(3):288-94. doi: 10.1111/j.1600-0838.2011.01398.x. Epub 2011 Nov 11. PMID 22092886
- [Background] Seminati E, Minetti AE. Overuse in volleyball training/practice: A review on shoulder and spine-related injuries. Eur J Sport Sci. 2013;13(6):732-43. doi: 10.1080/17461391.2013.773090. Epub 2013 Mar 5. PMID 24251752